CLINICAL TRIAL: NCT00663897
Title: A Comparative Study of Lansoprazole and Mosapride for Functional Dyspepsia: Focus on Difference Between Epigastric Pain Syndrome and Postprandial Distress Syndrome
Brief Title: Lansoprazole Versus Mosapride for Functional Dyspepsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lotung Poh-Ai Hospital (Other)
Collaborators: Tomorrow Medical Foundation (Other)
Responsible Party: Hsing-Hong Chen/Superintendent, Lotung Poh-Ai hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMCP-97-007
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Functional Dyspepsia; Epigastric Pain Syndrome; Post Prandial Distress Syndrome
Keywords: functional dyspepsia; epigastric pain syndrome; postprandial distress syndrome; proton pump inhibitor; 5 HT-4 receptor agonist
MeSH Terms: interventions — Lansoprazole; mosapride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Treatment with lansoprazole (30 mg) once daily for 14 days
  Interventions: Drug: lansoprazole
- 2 (Active Comparator): Treatment with mosapride (5 mg) thrice daily for 14 days
  Interventions: Drug: mosapride

INTERVENTIONS:
Drug: lansoprazole — lansoprazole, 30 mg, once daily for 14 days
  Other Names: Takepron (brand name)
  Arms: 1
Drug: mosapride — mosapride, 5 mg, thrice daily for 14 days
  Other Names: Mopride (brand name)
  Arms: 2

SUMMARY:
Functional dyspepsia is a common symptom complex with significant impact on quality of life. There is no standard treatment for functional dyspepsia but therapeutic efficacy of proton pump inhibitor (PPI) and prokinetic agent have been proved in subsets of patients. This study has two aims:

* first is to compare the therapeutic efficacy of lansoprazole (a PPI) and mosapride (a prokinetic agent) for functional dyspepsia
* second is to investigate whether different subgroups of functional dyspepsia (e.g., epigastric pain syndrome and postprandial distress syndrome) respond differently to PPI and prokinetic agent.

DETAILED DESCRIPTION:
Eligible outpatients with presentation of dyspepsia are enrolled if they fulfilled the criteria of ROME III criteria. A trained assistant helps the eligible patients to complete the ROME III standard questionaire, brief symptom rating scale (BSRS), and Maudsley Personality Inventory (MPI). The enrolled patients are then randomized into either lansoprazole or mosapride group for 14-day treatment. Before starting medication, right after completing the medication, and 1 month after the medication, the enrolled patients complete standardized severity questionnaire (Hong-Kong Index) to evaluate severity of dyspeptic symptoms. Symptom improvement is then determined.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 20 years old
* diagnosis of functional dyspepsia by fulfilling Rome-III criteria
* outpatient

Exclusion Criteria:

* aged less than 20 years
* organic lesions including ulcers, tumors, bleeding, vasculopathy or esophagitis as demonstrated on upper endoscopy
* concurrent illness with malignancy, diabetes mellitus, liver cirrhosis, renal failure or porphyria
* diagnosis of organic disease for dyspeptic symptoms by treating physicians
* history of abdominal surgery
* concurrent user of aspirin and NSAID
* history of allergy or severe side effects to lansoprazole or mosapride
* pregnant or lactating women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Improvement of dyspeptic symptoms as evaluated by validated questionnaire | After 2-week treatment of lansoprazole or mosapride

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Chun Hsu, M.D., Principal Investigator — Lotung Poh-Ai hospital, I-Lan County, Taiwan
Locations (1):
- Lotung Poh-Ai hospital, Lotung Town, Ilan County, Taiwan

REFERENCES:
- [Derived] Hsu YC, Liou JM, Yang TH, Hsu WL, Lin HJ, Wu HT, Lin JT, Wang HP, Wu MS. Proton pump inhibitor versus prokinetic therapy in patients with functional dyspepsia: is therapeutic response predicted by Rome III subgroups? J Gastroenterol. 2011 Feb;46(2):183-90. doi: 10.1007/s00535-010-0334-1. Epub 2010 Oct 19. PMID 20957498
- See also: The homepage of ROME foundation, an non-for-profit organization dedicated to scientific research and education information of functional gastrointestinal disorders (FGIDs). — http://www.romecriteria.org/